CLINICAL TRIAL: NCT05804864
Title: A Single-arm, Open, Multicenter Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Efficacy of the KM501 Double-antibody ADC in Subjects With Advanced Solid Tumors That Express, Amplify, or Mutate HER2
Brief Title: A Study of KM501 in Patients With Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM501-1001
Record Dates: First submitted 2023-03-12; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumors
Keywords: KM501; ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KM501-1001 (Experimental)
  Interventions: Drug: KM501

INTERVENTIONS:
Drug: KM501 — 1a: The program evaluated six dose levels, i.e., 0.1, 0.3, 0.6, 1.2, 1.8, 2.4 mg/kg, An accelerated titration was performed in the 0.1 and 0.3 mg/kg dose groups, and then a Bayesian optimal interval design was used to determine MTDS for four subsequent dose levels. Ib: The antitumor activity of KM501 monotherapy in subjects with specific types of tumors that are HER2-positive or express, amplify, or mutate will be evaluated at the RP2D dose level

SUMMARY:
A single-arm, open, multicenter Phase I study to evaluate the safety, tolerability, pharmacokinetic profile, and efficacy of the KM501 double-antibody ADC in subjects with advanced solid tumors that express, amplify, or mutate HER2

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent;
2. At least 18 years old and less than 75 years old on the date of signing the informed consent;
3. Subjects with histologically or cytologically confirmed advanced solid tumors who have developed disease progression since the last antitumor therapy, have no standard therapy available, do not tolerate or refuse standard therapy;

   * Stage Ia: Subjects with advanced relapsed or metastatic solid tumors with HER2 expression or amplification or mutation, stage Ia may refer to (but is not limited to) specific types of tumors at stage Ib;
   * Stage Ib: HER2-positive or expressed advanced breast cancer, advanced urothelial cancer, advanced gastric cancer or gastroesophageal junction adenocarcinoma, advanced ovarian cancer, and advanced endometrial cancer; Wild-type unresectable RAS and BRAF with HER2 expression or amplification in locally advanced or metastatic colorectal cancer; Advanced non-small cell lung cancer with a HER2 mutation. Other advanced tumors that are HER2-positive or expressed, HER2 amplified or mutated may be determined after discussion with the sponsor.
4. The subject shall provide a previous HER2 test report. If there is no previous HER2 test result, the archived/biopsied tumor tissue shall be provided for HER2 test in a 3A hospital or central laboratory. The HER2 status of the tumor tissue was determined by the investigator based on previous reports and test results from a 3A hospital or central laboratory. HER2 status is as follows:

   * HER2 expression: IHC(3+), IHC(2+) or IHC(+);
   * HER2 positive: IHC(3+) or IHC(2+) further test positive for ISH;
   * HER2 amplification: ISH positive or NGS/PCR confirmed HER2 amplification; • HER2 mutation: A HER2 mutation identified by NGS/PCR/Sanger sequencing.
5. The ECOG physical status score is 0 or 1 ;
6. Lesion requirements: Stage Ia subjects need to have evaluable lesions; Stage Ib subjects must have at least one measurable target lesion. For targets previously treated with radiation, a measurable lesion is considered only if there is definite progression [see Appendix 3 for the definition of measurable lesions in solid tumors].
7. Expected survival ≥12 weeks; 8. Within 7 days prior to initial drug administration, subjects must meet the following laboratory test values to ensure adequate organ and hematopoietic function (no blood transfusion, erythropoietin, granulocyte colony stimulating factor and other hematopoietic growth factor treatment, hepatoprotective therapy or other medical support treatment within 2 weeks prior to initial drug administration).

9. A man or woman with reproductive potential must consent to the use of effective contraceptive methods starting with the signing of an informed consent form and continuing for six months from the end of the study treatment (Appendix 6). Pregnancy tests for women of reproductive age must be negative within 7 days of the first trial drug administration (fertility potential defined as premenopausal women who have not had a tubal ligation or hysterectomy, or within 1 year after menopause).

Exclusion Criteria:

1. Subjects with known clinical or untreated central nervous system metastases, including meningeal metastases. Does not include: After radiation therapy, MRI/CT examination at least 4 weeks prior to initial administration of the trial drug (showing stable lesions, no uncontrollable neurological symptoms or signs (e.g., epilepsy, headache, central nausea/vomiting, progressive neurological dysfunction, papilledema), or any treatment that does not require local (e.g., radiation) and systemic (e.g., Untreated asymptomatic brain metastases of mannitol or corticosteroids;
2. Subjects with other malignancies within 5 years prior to initial administration of the experimental drug, except those with basal cell carcinoma, local squamous cell carcinoma of the skin, cervical carcinoma in situ, etc., who have not relapsed and metastasized after radical treatment;
3. Subjects who have received chemotherapy, targeted therapy, or other systematic antitumor therapy within 4 weeks or 5 half-lives (whichever is older) prior to the initial administration of the test drug, and who have been treated with Chinese herbal or proprietary drugs for antitumor purposes within 2 weeks prior to the initial administration;
4. Subjects who required systematic treatment with a dose of a corticosteroid >10 mg/ day equivalent to prednisone (see Appendix 9 for dose conversion) or other immunosuppressant within 14 days prior to initial administration of the trial drug or during the study period. Inhaled or topical doses ≤10 mg/ day equivalent to prednisone are permitted in the absence of active autoimmune disease. Short-term use of corticosteroids in doses >10 mg/ day equivalent to prednisone is permitted for the prevention (e.g., contrast allergy) or treatment of non-autoimmune diseases (e.g., delayed hypersensitivity caused by exposure to allergens);
5. Subjects who received major surgery (as determined by the investigator) or radical radiation therapy within 4 weeks prior to initial administration of the test drug; Or received palliative radiotherapy within 2 weeks prior to initial administration of the trial drug; Or received radioactive agents (strontium, samarium, etc.) for therapeutic purposes within 8 weeks prior to the first dosing of the test drug;
6. Subjects who have received other investigational drugs or treatments within 4 weeks prior to initial administration of the investigational drug;
7. ILD (non-infectious) interstitial lung disease (ILD) requiring glucocorticosteroid treatment/or current clinically significant active or current ILD/ pneumonia, or suspicious ILD/ pneumonia that cannot be excluded by imaging during screening;
8. Subjects with a known history of human immunodeficiency virus (HIV) infection; Laboratory test value: ANC≥ 1.5×109/L; PLT≥ 100×109/L Hb≥ 90 g/L ; CR≤1.5 times the upper limit of normal range (ULN) and creatinine clearance ≥60 mL/min (calculated according to Cockcroft-Gault formula); T-BIL ≤ 1.5 times ULN; ALT and AST Stage Ia: ≤ 2.5 times ULN;Stage Ib: ≤ 2.5 ULN, or ≤5 ULN (for subjects with liver metastases); INR and PT≤ 1.5 times ULN; APTT≤ 1.5 times ULN;
9. Active hepatitis B virus (HBsAg positive and/or HBcAb positive with HBV-DNA> upper limit of quantification) or hepatitis C virus infection (HCV antibody positive and HCV RNA positive);
10. Active infections requiring systematic treatment, including active tuberculosis, within 2 weeks prior to initial administration of the experimental drug;
11. Pleural effusion, pericardial effusion, and abdominal effusion that could not be controlled by appropriate intervention were present within 4 weeks prior to initial administration of the test drug (note: Subjects with small amounts of effusion that could only be detected by imaging examination could be included);
12. Subjects who have received previous organ transplants;
13. Toxicity associated with previous antitumor therapy did not return to grade 1 or less (NCI-CTCAE v5.0) (except for alopecia, grade 2 hypoparathyroidism, or toxicity judged by the investigator to be of no safety risk);
14. Subjects with active gastrointestinal bleeding, intestinal obstruction, intestinal paralysis, glaucoma, uncontrolled diabetes and other serious concomitant diseases;
15. Subjects with a known history of alcohol or drug abuse;
16. Subjects with significant cardiovascular disease: Subjects with severe arrhythmias, acute myocardial ischemia, unstable angina pectoris, congestive heart failure (NYHA grade ≥ 2 (Appendix 5)), left ventricular ejection fraction (LVEF) <50% within 6 months prior to initial administration of the experimental drug, Subjects with a history of long QT syndrome or a confirmed family history of long QT syndrome had heart-rate adjusted QTcF intervals of > 450 msec (male) and > 470 msec (female) using the Fridericia formula (Appendix 7);
17. Uncontrolled hypertension with standard treatment (systolic blood pressure ≥140 and/or diastolic blood pressure ≥90 mmHg);
18. History of cerebrovascular accidents, including transient ischemic attack or stroke, within 6 months prior to initial administration of the experimental drug;
19. Subjects with stage Ib colorectal cancer: subjects with known activating mutations in exons 2, 3, and 4 of KRAS/NRAS and V600E of BRAF (except those who are assessed to benefit by the investigator);
20. Subjects with a history of grade 2 or above peripheral nerve disease;
21. People who are known to be allergic to recombinant humanized anti-HER-2 bispecific antibody -MMAE conjugate drug and its components (L-histidine, histidine hydrochloride, polysorbate 80, etc.);
22. Previous history of hypersensitivity, angioedema or severe hypotension caused by Herceptin or pertuzumab or biosimilar drugs;
23. Subjects with a known mental illness that may affect compliance with the test;
24. Pregnant women (positive pregnancy test before medication) or lactating women;
25. The investigator considers that the subject is ineligible to participate in the clinical study for any clinical or laboratory abnormality or other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (for Part 1a) | Up to 4weeks
  Determine MTD of KM501
Recommended phase 2 dose (RP2D) (if has) (Part 1a) | Up to 4 weeks.
  Determine Recommended Phase 2 dose (RP2D) of KM501
Number of participants with treatment-related adverse events （Part 1a） | Up to 8 months.
  Incidence of AE as assessed by CTCAE 5.0
Objective response rate (ORR) (Part 1b) | Up to 2-3 years.
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Area under the concentration versus time curve of KM501 in plasma (AUC)(Part 1a and Part1b). | Up to 8 months for Part 1a; Up to 2 to 3 years for Part1b.
  To determine the area under the plasma concentration time curve (AUC) of KM501
Maximum plasma concentration (Cmax) of KM501(Part 1a and Part 1b ). | Up to 63days for Part 1a; Up to 63 days for Part1b.
  Cmax is the maximum observed plasma concentration in ng/mL
Serum Half-life (T-HALF) of KM501. (Part1a and Part1b) | Up to 63days.
  To determine the t1/2 of KM501.
Anti-drug antibody(ADA )OF KM501 . (Part1a and Part1b) | up to 8months for Part1a and up to 2-3 years for Part1b.
  To determine the immunogenicity of KM501.
Objective response rate (ORR) (Part 1a) | Up to 8months.
  Number of participants who achieved a best response of either complete response (CR) or partial response (PR) during treatment evaluated by investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression free survival (PFS) (Part 1a and Part 1b) | up to 2-3 years.
  To determine the PFS by investigator.
Disease control rate (DCR) (Part 1a and Part 1b) | up to 2-3 years.
  To determine the DCR by investigator.
Overall survival (OS) (Part1a and Part1b ) | up to 2-3 years
  To determine the OS by investigator.
Number of patients with adverse events (Part 1b) | up to 2-3 years.
  Incidence of AE as assessed by CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China